CLINICAL TRIAL: NCT00100464
Title: Serotonin and the Upper Airway in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RESP-013-98F
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Serotonin; Sleep Apnea Syndrome; Pharyngeal Muscles
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Paroxetine

INTERVENTIONS:
Drug: Paroxetine
Drug: 5HTP

SUMMARY:
The purpose of this study is to determine if a certain medication, alone or combined with another medication, will increase muscle activity in the upper airway in people who do and people who do not have sleep apnea. The medications being studied are paroxetine, a commonly used antidepressant, and 5 hydroxy-tryptophan (5HTP), which also can be used as a dietary supplement without a prescription. Because the effects of paroxetine in previous studies were not very large, we will also study it combined with 5HTP to see if the effect on the upper airway muscles is greater.

ELIGIBILITY:
Group A: 20 Adult patients with mild to severe sleep apnea. If patients are being treated with nasal CPAP, they will continue treatment except on study nights.

Group B: 20 normal adult non-snoring subjects.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 2000-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Malcolm Randall VA Medical Center, Gainesville, Florida, United States